CLINICAL TRIAL: NCT07097974
Title: Evaluation of the Efficacy of the Composite WM Formula in Body Weight Change
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 25-047-A
Record Dates: First submitted 2025-07-30; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Obesity
Keywords: Probiotic; Prebiotic; Glucagon-like peptide-1 (GLP-1); Blood glucose; Insulin
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WM formula liquid drink (Experimental): WM formula liquid drink, 50 g/glass jar
  Interventions: Dietary Supplement: WM formula liquid drink
- Placebo (Placebo Comparator): The placebo contained the same base ingredients as the WM formula but without the active WM formula component.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: WM formula liquid drink — One glass jar (50 g) of the WM formula liquid drink was administered once daily, 1 hour prior to the first meal of the day.
  Arms: WM formula liquid drink
Dietary Supplement: Placebo — One glass jar (50 g) of the placebo liquid drink was administered once daily, 1 hour prior to the first meal of the day.
  Arms: Placebo

SUMMARY:
This study aims to evaluate the effects of the combined formula WM Formula, used as a dietary supplement, with a focus on improvements in glycemic and lipid parameters, body composition, and gut microbiota profiles.

DETAILED DESCRIPTION:
This study is a single-center, randomized, double-blind, placebo-controlled human clinical trial designed to evaluate the potential effect of the WM Formula composite supplement on body weight. Eligible participants will be adults aged 18 years or older, screened based on waist circumference or body fat percentage.

Participants will be randomly assigned to one of two groups: one receiving the combined formula WM Formula, and the other receiving a placebo. Each group will take either the WM Formula or placebo, and undergo regular assessments throughout the 4-week study period. Physiological parameters (e.g., height, weight, blood pressure, BMI) and biochemical markers (including liver and kidney function, lipid profile, and blood glucose levels) will be collected at baseline (Week 0), Week 2, and Week 4. In addition, participants will complete appetite assessment questionnaires and other surveys to evaluate changes in appetite and gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older who are willing to sign the informed consent form.
* Body fat percentage: ≥30% for females and ≥25% for males.
* Non-pregnant and non-lactating women who agree to use physical contraceptive methods (e.g., condoms, intrauterine devices) throughout the study period.

Exclusion Criteria:

* Use of GLP-1 receptor agonists approved in Taiwan (e.g., liraglutide, semaglutide, dulaglutide), blood glucose-regulating medications, weight loss-related drugs or functional foods, probiotics, or gastrointestinal health-related supplements or medications within 30 days prior to the start of the study.
* History of chronic gastrointestinal disorders, seizure disorders or epilepsy, hepatic or renal diseases, malignancies, endocrine disorders, psychiatric illnesses, alcohol or drug abuse, or other major organic diseases based on medical history.
* History of gastrointestinal surgery, organ transplantation, or other major surgeries.
* History of hypoglycemia.
* Known lactose intolerance.
* Chronic diarrhea.
* Acute gastroenteritis within 2 weeks prior to study initiation.
* Known allergy to any ingredient in the investigational product.
* Employees or immediate family members of TCI Co., Ltd.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in weight at weeks 2 and 4 | Week 0, 2 and 4
  Assessment of changes in weight at baseline, week 2, and week 4
Change from plasma GLP-1 concentration (pmol/L) in baseline at weeks 2 and 4 | Assessment of changes in GLP-1 concentration at baseline, week 2, and week 4
Change from baseline in blood glucose at weeks 2 and 4 | Week 0, 2 and 4
  Assessment of blood glucose changes at weeks 0, 2, and 4

SECONDARY OUTCOMES:
Change from plasma DPP-4 concentration (ng/mL) in baseline at weeks 2 and 4 | Week 0, 2 and 4
  Assessment of plasma DPP-4 concentration changes at weeks 0, 2, and 4
Change from plasma PAI-1 concentration (ng/mL) in baseline at weeks 2 and 4 | Week 0, 2 and 4
  Assessment of plasma PAI-1 concentration changes at weeks 0, 2, and 4

CONTACTS AND LOCATIONS:
Locations (1):
- TCI Co., Ltd., Taipei, Taiwan